CLINICAL TRIAL: NCT01828177
Title: A Multicenter Randomized Evaluator-Blinded Vehicle-Controlled Parallel Group Evaluation of Twice Daily PDI-320 in Comparison to Its Monads in Adults With Rosacea
Brief Title: An Evaluation of PDI-320 in Comparison to Its Monads in Adults With Rosacea
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PreCision Dermatology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 172-7451-201
Record Dates: First submitted 2013-04-03; First posted 2013-04-10 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Rosacea
Keywords: PreCision; PDI-320; Foam
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PDI-320 (Experimental): Foam, twice daily for up to 12 weeks
  Interventions: Drug: PDI-320
- PDI-320 Monad #1 (Experimental): Foam, twice daily for up to 12 weeks
  Interventions: Drug: PDI-320 Monad #1
- PDI-320 Monad #2 (Experimental): Foam, twice daily for up to 12 weeks
  Interventions: Drug: PDI-320 Monad #2
- Vehicle (Placebo Comparator): Foam, twice daily for up to 12 weeks
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: PDI-320
  Arms: PDI-320
Drug: PDI-320 Monad #1
  Arms: PDI-320 Monad #1
Drug: PDI-320 Monad #2
  Arms: PDI-320 Monad #2
Drug: Vehicle
  Arms: Vehicle

SUMMARY:
This 4-arm Phase 2 vehicle-controlled study is designed to assess the safety and efficacy of PDI-320, and the individual components, in adult subjects with rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Subject has moderate to severe papulopustular rosacea and at least mild erythema and mild telangiectasia.
* Subject is willing and able to apply the test article(s) as directed, comply with study instructions and commit to all follow-up visits for the duration of the study.
* If subject is a woman of childbearing potential, she must have a negative urine pregnancy test and agree to use an effective form of birth control for the duration of the study.

Exclusion Criteria:

* Subject is pregnant, lactating or is planning to become pregnant during the study.
* Subject has any other active dermatological condition on the face that may interfere with the conduct of the study.
* Subject has used systemic immunosuppressants within 30 days prior to study start.
* Subject has used systemic retinoids within 6 months prior to study start.
* Subject has used any topical rosacea therapy within 14 days prior to study start.
* Subject has had laser or light therapy on the face within 3 months of study start.
* Subject is currently enrolled in an investigational drug or device study.
* Subject has used an investigational drug or investigational device treatment within 30 days prior to first application of the test article.
* Subject has used vasodilators or adrenergic blocking agents within 6 weeks of study start (except subjects on stable dose for greater than 3 months).
* Subject has active ocular rosacea and/or blepharitis/meibomianitis requiring treatment by an ophthalmologist.
* Subject has previously failed to have improvement of rosacea with appropriate use of systemic tetracycline family of antibiotics or use of the components of PDI-320.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Treatment "Success Rate" based on change in Investigator's Global Assessment (IGA) | Baseline and End of Treatment (up to 12 weeks)
  IGA Score Success Rate is defined as the percentage of subjects who achieve "Clear" (score = 0) or "Almost Clear" (score = 1) and have at least a 2-grade improvement on the IGA score at the End of Treatment. IGA score is used to evaluate the overall severity of rosacea using a 5-point scale from 0 (clear) to 4 (severe).
Absolute change in inflammatory lesion count | Baseline and End of Treatment (up to 12 weeks)
  Inflammatory lesions include papules and pustules on the face, and are counted by study personnel.

SECONDARY OUTCOMES:
Treatment "Success Rate" based on change in IGA (interim time points) | Baseline, Week 4 and Week 8
  IGA Score Success Rate is the same as defined in the Primary Outcome Measures.
Absolute change in inflammatory lesion count (interim time points) | Baseline, Week 4 and Week 8
  Inflammatory lesions include papules and pustules on the face, and are counted by study personnel.
Change in erythema severity | Baseline and End of Treatment (up to 12 weeks)
  The investigator will assess the erythema (skin redness) on the entire face, using a grading scale from 0 (none) to 4 (very severe)
Change in telangiectasia severity | Baseline and End of Treatment (up to 12 weeks)
  The investigator will assess telangiectasia (small dilated blood vessels near the surface of the skin) on the face, using a grading scale of 0 (none) to 3 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Syd Dromgoole, PhD, Study Director — Therapeutics, Inc.
Locations (2):
- United States (2):
  - Therapeutics Clinical Research, San Diego, California
  - Academic Dermatology Associates, Albuquerque, New Mexico